CLINICAL TRIAL: NCT02400749
Title: A Double-blind, Placebo-controlled, Randomized Study on the Safety and Efficacy of Apremilast in Patients With Moderate to Severe Plaque Psoriasis Involving Palms and/or Soles
Brief Title: Apremilast in Palmo-Plantar Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Inno-6040; AP-CL-PSOR-CARE-005313 (Other: Celgene)
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Results first posted 2018-10-24 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-10

CONDITIONS: Palmo-plantar Psoriasis
Keywords: moderate to severe non-pustular palmo-plantar psoriasis
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apremilast (Experimental): Patients will receive Apremilast until week 32.
  Interventions: Drug: Apremilast
- Placebo followed by Apremilast (Placebo Comparator): Patients will receive Placebo until week 16 and then receive Apremilast until week 32
  Interventions: Drug: Apremilast; Drug: Placebo

INTERVENTIONS:
Drug: Apremilast — Apremilast tablets will be provided to sites in blister cards.
  Patients will be provided a titration blister pack containing apremilast 10 mg, 20 mg and 30 mg at the Day 0 and week 16 visits (refer to section 6.1). Following the 6 day titration period (for Day 0 and week 16) blister packs will contain apremilast 30 mg bid or placebo bid.
  Other Names: OTEZLA
Drug: Placebo — Placebo tablets will be provided to sites in blister cards.
  Arms: Placebo followed by Apremilast

SUMMARY:
This study will compare the safety and efficacy of Apremilast 30mg to placebo in subjects with moderate to severe plaque psoriasis involving palms and/or soles.

Apremilast will be administered orally twice daily for 16 to 32 weeks, and will be compared against placebo (dummy drug with no active ingredient).

This study will enroll approximately 100 adult subjects with moderate to severe plaque psoriasis involving palms and/or soles in approximately 20 centers in US and Canada. To be eligible, subjects must have moderate to severe plaque psoriasis involving palms or soles, with lesions covering at least 10% of the surface of palms and soles at the baseline visit. Study treatments will be assigned randomly (like flipping a coin) at a 1:1 ratio, meaning that there will be a 1 in 2 chance of either receiving Apremilast or placebo during the first 16 weeks. Subjects will not know which of the two treatments they receive. The study doctor, the study staff will not know which treatment they receive either. All subjects will receive Apremilast from Week 16 to Week 32.

Subjects will be asked to complete questionnaires about their hand and feet pain, their quality of life, their general health and the impact of psoriasis on their work.

Medical photographs of palms and soles will be taken for subjects at selected study sites only.

At Baseline and Week 16 visits, for willing subjects at certain study sites, skin biopsies can be taken. The biopsies will be analyzed for the presence of antibodies, antigens or certain cellular messengers that can be quantified. It is also possible to study the skin cellular structure and organization.

A total of 3 biopsies will be taken: At Baseline visit, one biopsy from psoriasis on palms or soles and one biopsy from normal skin of palms or soles will be collected. At Week 16 visit, only one biopsy from psoriasis on palms or soles will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Patient, male or female, is aged 18 years or older at the screening visit.
2. Patient has a history of plaque psoriasis involving the palm(s) and/or sole(s) for at least 6 month(s).
3. Patient has moderate to severe psoriasis with a PPPGA of at least 3 and with at least 10% of the total surface of palms and soles (PPPSA) affected by psoriatic plaques at baseline.

Exclusion Criteria:

1. Female patient is pregnant or breastfeeding
2. Patient has the presence of pustules on palms or soles at screening or baseline
3. Patient who has used any topical treatment for psoriasis (except non-medicated emollients) in the last 14 days before Day 0 with the exception of hydrocortisone and desonide for the face, groin (including genitals) and inframammary areas as well as shampoos containing tar, salicylic acid or zinc pyrithione if they are applied with gloves.
4. Patient who has used ultraviolet B (UVB) phototherapy or excessive sun exposure less than 28 days before Day 0.
5. Patient has used any non-biological systemic therapy for the treatment of psoriasis (including psoralens ultraviolet A (PUVA)) therapy, methotrexate, acitretin and cyclosporin), systemic steroids or systemic immunosuppressants less than 28 days before Day 0.
6. Use of any investigational agents within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamic half-lives, if known (whichever is longer).
7. Prior treatment with apremilast
8. Patient is currently participating in a clinical trial with an experimental agent or device.
9. Patient is using or has used any biological therapy for the treatment of psoriasis. Exceptions to this criterion are: patients who used no more than one biologic in the past and stopped for reasons other than lack of efficacy are eligible.
10. Patient is taking or requires oral or injectable corticosteroids during the study. Inhaled corticosteroids for stable medical conditions are allowed. Patients who have used oral or injectable corticosteroids less than 28 days before Day 0 are excluded.
11. Patient is known to have immune deficiency or is immunocompromised or currently uses or plans to use anti-retroviral therapy at any time during the study.
12. Active tuberculosis or history of inadequately treated tuberculosis
13. Other than psoriasis, patient has any clinically significant (as determined by the Investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is currently uncontrolled.
14. Other than psoriasis, patient has any other dermatological condition that could, in the opinion of the investigator, interfere with the study assessments.
15. Any condition, including the presence of laboratory abnormalities (including estimated creatinine clearance of less than 30 mL per minute), which would place the patient at unacceptable risk if he/she were to participate in the study.
16. Malignancy or history of malignancy, except for:

    * treated [ie, cured] basal cell or squamous cell in situ skin carcinomas;
    * treated [ie, cured] malignancy with no evidence of recurrence within the previous 5 years.
17. Known hypersensitivity to apremilast or any excipients in formulation.
18. Patient has the following hereditary disease: galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
19. Use of strong cytochrome P450 enzyme inducers (e.g. rifampin, phenobarbital, carbamazepine, phenytoin)
20. Active substance abuse or a history of substance abuse within 6 months prior to Screening.
21. Prior history of suicide attempt at any time in the patient's life time prior to screening or randomization, or major psychiatric illness requiring hospitalization within the last 3 years.
22. Presence of uncontrolled depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, FRCPC, Principal Investigator — Innovaderm Research Inc.
Locations (11):
- Innovaderm Investigational Site, Arlington Heights, Illinois, United States
- Canada (10):
  - Innovaderm Investigational Site, Calgary, Alberta
  - Innovaderm Investigational Site, St. John's, Newfoundland and Labrador
  - Innovaderm Investigational Site, Barrie, Ontario
  - Innovaderm Investigational Site, Markham, Ontario
  - Innovaderm Investigational Site, North Bay, Ontario
  - Innovaderm Investigational Site, Peterborough, Ontario
  - Innovaderm Investigational Site, Drummondville, Quebec
  - Innovaderm Investigational Site, Montreal, Quebec
  - Innovaderm Investigational Site, Saint-Jérôme, Quebec
  - Innovaderm Investigational Site, Québec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Apremilast: Patients will receive apremilast until Week 32.
  Apremilast: Apremilast tablets provided to sites in blister cards.
  Patients will be provided a titration blister pack containing apremilast 10 mg, 20 mg and 30 mg at Day 0 and Week 16 visits. Following a 6-day titration period (for Day 0 and Week 16), patients will use blister packs containing apremilast 30 mg bid.
- Placebo Followed by Apremilast: Patients will receive Placebo until Week 16 and then receive apremilast until Week 32
  Placebo/Apremilast: Placebo and apremilast tablets provided to sites in blister cards.
  Patients will be provided a titration blister pack containing placebo at the Day 0 visit and apremilast 10 mg, 20 mg and 30 mg at the Week 16 visit (refer to section 6.1). Following the 6 day titration period (for Day 0 and Week 16), patients will receive blister packs containing apremilast 30 mg bid or placebo bid.
Period: Week 0 -16
Arm/Group | Apremilast | Placebo Followed by Apremilast
Started | 50 | 50
Completed | 39 | 44
Not Completed | 11 | 6
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 1 | 0
Period: Week 17 - 32
Arm/Group | Apremilast | Placebo Followed by Apremilast
Started | 39 | 44
Completed | 34 | 41
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apremilast | Placebo Followed by Apremilast | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (8.6) | 53.6 (13.5) | 55.1 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 59
  Male | 20 | 21 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 3 | 6
  Black | 1 | 0 | 1
  Caucasian | 45 | 47 | 92
  Other | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 50 | 50 | 100
Smoking Status [Count of Participants; unit: Participants]
  Never | 12 | 19 | 31
  Past | 18 | 18 | 36
  Present | 20 | 13 | 33
Weight [Mean (Standard Deviation); unit: kg] | 86.9 (17.1) | 88.3 (19.8) | 87.6 (18.4)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.1 (5.5) | 31.0 (6.6) | 31.0 (6.0)
Palmoplantar Psoriasis Physician Global Assessment (PPPGA) [Count of Participants; unit: Participants] — The PPPGA is a zero to five, 6-point scale that evaluates the severity of palmoplantar psoriasis (score 0 [Clear]; score 1 [Almost clear]; score 2 [Mild]; score 3 [Moderate]; score 4 [Severe]; score 5 [Very severe]).
  Participants
    Score 3 | 30 | 32 | 62
    Score 4 | 19 | 16 | 35
    Score 5 | 1 | 2 | 3
Palmoplantar Psoriasis Physician Global Assessment (PPPGA) [Mean (Standard Deviation); unit: units on a scale] — The PPPGA is a zero to five, 6-point scale that evaluates the severity of palmoplantar psoriasis (score 0 [Clear]; score 1 [Almost clear]; score 2 [Mild]; score 3 [Moderate]; score 4 [Severe]; score 5 [Very severe]).
  units on a scale | 3.4 (0.5) | 3.4 (0.6) | 3.4 (0.6)
Palmoplantar Psoriasis Area Severity Index (PPPASI) [Mean (Standard Deviation); unit: units on a scale] — The PPPASI is a scale that can vary from 0 to 72.
  Erythema (E), induration (I), and desquamation (D) are evaluated on a scale of 0 to 4 while area is evaluated on a scale of 0 to 6. The combined score of each of these features, for the right (R) and left (L) palms and soles, gives a PPPASI score from 0 (absence of disease) to 72 (most severe palmoplantar psoriasis possible).
  PPPASI = (E + I + D)Area X 0.2 (R palm) + (E + I + D) Area X 0.2 (L palm) + (E + I + D) Area X 0.3 (R sole) + (E + I + D) Area X 0.3 (L sole)
  units on a scale | 18.7 (11.3) | 15.6 (8.5) | 17.1 (10.1)
Palmoplantar Psoriasis Surface Area (PPPSA) [Mean (Standard Deviation); unit: units on a scale] — The surface affected by psoriasis on palms and soles is estimated as a percentage of the total surface of palms and soles. Each palm represents 20% and each sole 30%. PPPSA values range from 0% (no psoriasis on palms and soles) to 100% (all palms and soles covered by psoriasis).
  units on a scale | 38.1 (23.4) | 30.5 (18.3) | 34.3 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: Palmoplantar Psoriasis Physician Global Assessment (PPPGA) of 0 or 1
Description: Number of patients who achieve a PPPGA of 0 or 1 at Week 16 for patients randomized to apremilast as compared to patients randomized to placebo
  The PPPGA is a zero to five, 6-point scale that evaluates the severity of palmoplantar psoriasis (score 0 [Clear]; score 1 [Almost clear]; score 2 [Mild]; score 3 [Moderate]; score 4 [Severe]; score 5 [Very severe]).
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast | Placebo Followed by Apremilast
Number analyzed (Participants) | 50 | 50
Participants | 7 | 2

2. Secondary Outcome: Palmoplantar Psoriasis Physician Global Assessment (PPPGA)
Description: Change from baseline in mean PPPGA at Week 16 for patients randomized to apremilast as compared to patients randomized to placebo
  The PPPGA is a zero to five, 6-point scale that evaluates the severity of palmoplantar psoriasis (score 0 [Clear]; score 1 [Almost clear]; score 2 [Mild]; score 3 [Moderate]; score 4 [Severe]; score 5 [Very severe]).
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast | Placebo Followed by Apremilast
Number analyzed (Participants) | 50 | 50
units on a scale | -0.8 (1.0) | -0.4 (0.8)

3. Secondary Outcome: Palmoplantar Psoriasis Area Severity Index (PPPASI)
Description: Change from baseline in PPPASI at Week 16 for patients randomized to apremilast as compared to patients randomized to placebo
  Palmoplantar psoriasis area severity index (PPPASI) is a scale that can vary from 0 to 72.
  Erythema (E), induration (I), and desquamation (D) are evaluated on a scale of 0 to 4 while area is evaluated on a scale of 0 to 6. The combined score of each of these features, for the right (R) and left (L) palms and soles, gives a PPPASI score from 0 (absence of disease) to 72 (most severe palmoplantar psoriasis possible).
  PPPASI = (E + I + D)Area X 0.2 (R palm) + (E + I + D) Area X 0.2 (L palm) + (E + I + D) Area X 0.3 (R sole) + (E + I + D) Area X 0.3 (L sole)
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast | Placebo Followed by Apremilast
Number analyzed (Participants) | 50 | 50
units on a scale | -7.4 (7.1) | -3.6 (5.9)

4. Secondary Outcome: Palmoplantar Psoriasis Surface Area (PPPSA)
Description: Change from baseline in PPPSA at Week 16 for patients randomized to apremilast as compared to patients randomized to placebo
  The surface affected by psoriasis on palms and soles is estimated as a percentage of the total surface of palms and soles. Each palm represents 20% and each sole 30%. PPPSA values range from 0% (no psoriasis on palms and soles) to 100% (all palms and soles covered by psoriasis).
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast | Placebo Followed by Apremilast
Number analyzed (Participants) | 50 | 50
units on a scale | -0.1 (0.1) | 0.0 (0.2)

5. Secondary Outcome: Palmoplantar Psoriasis Area Severity Index (PPPASI)
Description: Change from baseline in PPPASI at Week 32 for patients randomized to apremilast
  Palmoplantar psoriasis area severity index (PPPASI) is a scale that can vary from 0 to 72.
  Erythema (E), induration (I), and desquamation (D) are evaluated on a scale of 0 to 4 while area is evaluated on a scale of 0 to 6. The combined score of each of these features, for the right (R) and left (L) palms and soles, gives a PPPASI score from 0 (absence of disease) to 72 (most severe palmoplantar psoriasis possible).
  PPPASI = (E + I + D)Area X 0.2 (R palm) + (E + I + D) Area X 0.2 (L palm) + (E + I + D) Area X 0.3 (R sole) + (E + I + D) Area X 0.3 (L sole)
Time Frame: 32 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 50
units on a scale | -11.3 [-14.1 to -8.5]

6. Secondary Outcome: Palmoplantar Pustulosis Physician Global Assessment (PPPGA) of 0 or 1
Description: Number of patients who achieve a PPPGA of 0 or 1 at Week 32 for patients randomized to apremilast
  The PPPGA is a zero to five, 6-point scale that evaluates the severity of palmoplantar psoriasis (score 0 [Clear]; score 1 [Almost clear]; score 2 [Mild]; score 3 [Moderate]; score 4 [Severe]; score 5 [Very severe]).
Time Frame: 32 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast
Number analyzed (Participants) | 50
Participants | 12

ADVERSE EVENTS:
Time Frame: After the first study drug administration and until the end of study at Week 32.
Arm/Group | Apremilast | Placebo Followed by Apremilast
Serious Adverse Events (participants affected / at risk) | 3/50 | 2/50
Other Adverse Events (participants affected / at risk) | 27/50 | 29/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apremilast (N=50) | Placebo Followed by Apremilast (N=50)
myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
breast cancer requiring hospitalization for bilateral mastectomy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
E. coli bacteremia, C-difficile + hypokalemia requiring hospitalization (Infections and infestations) | 1 (1) | 0 (0)
carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apremilast (N=50) | Placebo Followed by Apremilast (N=50)
Diarrhoea (Gastrointestinal disorders) | 9 (13) | 9 (15)
Frequent bowel movements (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (6) | 6 (6)
Fatigue (General disorders) | 3 (3) | 2 (2)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (6) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (8)
Headache (Nervous system disorders) | 8 (10) | 7 (8)

LIMITATIONS AND CAVEATS:
Clinical evaluations of psoriasis on palms and soles are not easy to perform. This is especially difficult for soles where frictional hyperkeratosis and physiological erythema is often difficult to differentiate form psoriasis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator have an obligation to present or publish the results in accordance with GCP, ICH, and the declaration of Helsinki, provided that confidential information and/or proprietary information of the sponsor, not publicly known is not disclosed without prior, written permission from the sponsor.